CLINICAL TRIAL: NCT03734406
Title: Can Video Clips Improve Patient Comprehension at the Emergency Department? A Multicentric Randomized Controlled Trial.
Brief Title: Can Video Clips Improve Patient Comprehension at the Emergency Department?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Santi Di Pietro, Clinical Research Coordinator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20180068344
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Doctor Patient Communication; Patient Safety; New Technologies in Clinical Medicine; Patient Education and Health Literacy; Safe Hospital Discharge

STUDY DESIGN:
Intervention Model Description: We designed a multicentric, pragmatic, parallel groups trial, with 1:1 randomization, that will involve patients discharged from EDs with a diagnosis of atrial fibrillation (AF) or deep vein thrombosis (DVT).
  The study aims to demonstrate the superiority of the intervention in terms of patients' comprehension of their medical condition, assessed with a telephone interview that will be conducted within 48 hours from patients' discharge.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): All subjects enrolled in the study group will be showed during the discharge process the video related to patient's condition (DVT vs AF), using it as a graphic support to doctor's verbal explanation of the diagnosed pathology and its possible complications.
  For the purposes of the study we have selected two 3D videoclips, available on various internet sites and not covered by any copyright restrictions; these have been modified and shortened to make them suitable to use in our study setting.
  The images contained show the pathophysiological process underlying the two diseases under study, namely deep vein thrombosis and atrial fibrillation.
  The SIs will show the videos to patients on the institutional computer or, alternatively, on their personal smartphone / tablet. The videos were purposely left without audio content.
  Interventions: Other: Videoclips
- Control group (No Intervention): Patients of the control group will receive discharge explanations without the aid of any video.
  The communication strategy in these cases won't be standardized, in order to leave the treating doctors free to express themselves in the way they are used to in their clinical practice, which is based solely on doctor's verbal and non-verbal communication skills.

INTERVENTIONS:
Other: Videoclips — The images contained in the videoclips show the pathophysiological process underlying the two diseases under study, namely deep vein thrombosis and atrial fibrillation.
  Arms: Video group

SUMMARY:
The aim of this study is to assess the utility of two interventional videos, showed to patients discharged from the ED with a diagnosis of atrial fibrillation or deep vein thrombosis. We have focused our attention on these two medical conditions because they share some important features: they are frequently seen in EDs; their main complication (stroke and pulmonary embolism) can cause significant morbidity and mortality; both conditions and their related complications are probably not very intuitive to comprehend for the general population. In fact, the understanding of these conditions implies the knowledge of a number of pathological processes, with which most people are unfamiliar.

The primary hypothesis is that patients enrolled in the study group will show a higher degree of comprehension of their medical condition and its related complications, as compared to the control group. Secondly, we will also analyze any possible effect of the videos on the knowledge of the therapy prescribed, return instructions and patients' satisfaction with the quality of communication in the ED.

Eventually, we will examine the association of some factors with the outcomes (age, sex, level of education, atrial fibrillation vs. deep vein thrombosis group).

ELIGIBILITY:
* Age >18
* Being diagnosed with one of the two medical condition under study: patients with first-time diagnosis of deep vein thrombosis; patients with first-time diagnosis of atrial fibrillation; patients with second episode in life of atrial fibrillation who have never been prescribed take-home medications for its cure or prevention of recurrence (anticoagulants, antiarrhythmic drugs including beta-blockers)
* Being discharged home directly from the Emergency Department/Emergency Unit
* Capacity of the patient to understand the explanations and instructions provided by the doctor (this includes excellent command of the Italian language)
* Having provided a valid phone number
* Having signed the informed consent

In case of patients lacking capacity, and in all cases of patients who will be judged by the recruiting doctor as incapable to safely receive the discharge instructions, the caregiver will be enrolled to the study with identical modalities.

In the context of a pragmatic trial, we did not set exclusion criteria in terms of education level and comorbidities of the enrolled patients.

Exclusion criteria:

* Previous diagnosis of deep vein thrombosis
* Two or more previous episodes of atrial fibrillation; or one previous episode of atrial fibrillation for which the patient has been prescribed one of the following take-home medications: anticoagulants, antiarrhythmic drugs including beta-blockers.
* Being hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Patient's comprehension of their medical condition and its potential complications | Outcome assessed within 48 hours from ED discharge
  The main outcome corresponds to interview's questions n°1-3-4. Patients' answers will receive a score on a 4-points Likert scale (from zero to three) from low to high knowledge.
  Scores from the two independent reviewers will be averaged and then added to obtain an overall score. The score for the main outcomes will therefore range 0-18 for the main outcome.
  To the best of our knowledge, no currently available validated questionnaires would serve for the purpose of our study, i.e. for the simultaneous measurement of different domains of comprehension across two different medical conditions.
  Hence, we have developed the ad-hoc interview and its related interpretation scheme using face and content validity. Construct validation would require an amount of time and resources equivalent to that of the trial itself, pushing it beyond practical feasibility.

SECONDARY OUTCOMES:
Patient's knowledge of the prescribed therapy | Outcome assessed within 48 hours from ED discharge
  This outcome is measured with interview's question n°2. Scores will range from 0-6 (low to high comprehension).
Patient's satisfaction | Outcome assessed within 48 hours from ED discharge
  This outcome is measured with interview's question n°5 and n°6. Scores will range from 0-12.

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department, IRCCS San Matteo University Hospital, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Pietro S, Ferrari I, Bulgari G, Muiesan ML, Falaschi F, De Silvestri A, Scudeller L, Musella V, Saglio S, Re B, Mattiuzzo E, Cherubini F, Perlini S; Improving Emergency Department Discharge Research Group. Video clips for patient comprehension of atrial fibrillation and deep vein thrombosis in emergency care. A randomised clinical trial. NPJ Digit Med. 2024 Apr 30;7(1):107. doi: 10.1038/s41746-024-01107-7. PMID 38688958